CLINICAL TRIAL: NCT00406744
Title: Evaluation of Efficacy of Intravitreal Bevacizumab Retreatments
Brief Title: Efficacy of Retreatments With Intravitreal Bevacizumab
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-0012
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Age Related Macular Degeneration; Choroidal Neovascularization
Keywords: neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization; Neovascularization, Pathologic

INTERVENTIONS:
Drug: Intravitreal injection of Bevacizumab

SUMMARY:
Choroidal neovascularization is a leading cause of visual loss in people older than 60 years and for its treatment there had been performed multicentric studies with Lucentis (Ranibizumab) with a significant improval of visual acuity. In our institution we evaluated efficacy of bevacizumab in several pathologies but we dont know what would be the results if we use the same dose several times. Our purpose was to determine the efficacy of bevacizumab for improve or stabilize visual acuity with two or more intravitreal inyections of bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* * Any visual acuity

  * OCT: Central foveal thickness greater than 300 u or with evidence of subretinal fluid.
  * Active angiogram leakage

Exclusion Criteria:

* * Basal Inflammatory disease

  * Endoftalmitis history
  * Lesions bigger than 5400 u or with scarring greater than 50% of lesion.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2006-05 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity, OCT foveal thickness and fluorescein angiogram

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Kon-Jara, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico, Mexico City, Mexico City, Mexico